CLINICAL TRIAL: NCT00377572
Title: Inner-City Anti-IgE Therapy for Asthma (ICAC-08)
Brief Title: Inner-City Anti-IgE Therapy for Asthma
Acronym: ICATA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Inner-City Asthma Consortium (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DAIT ICAC-08; ICATA (Other: NIAID)
Record Dates: First submitted 2006-09-14; First posted 2006-09-18 (Estimated); Results first posted 2013-06-07 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-02

CONDITIONS: Asthma
Keywords: Immunoglobulins; Immunoglobulin E; omalizumab; anti-IgE
MeSH Terms: conditions — Asthma | interventions — Omalizumab; anti-IgE antibodies

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Omalizumab (Xolair) + Conventional Therapy (Experimental): Omalizumab was administered subcutaneously every 2 or 4 weeks over a period of 60 weeks to participants classified as having moderate to severe asthma. Doses (mg) and dosing frequency were determined by serum total IgE level (IU/mL) and body weight (kg). Also, participants continued with their conventional asthma therapy according to the National Asthma Education and Prevention Program (NAEPP-II, 2002) guidelines, under the management of an asthma specialist health care provider.
  Interventions: Biological: omalizumab
- Placebo + Conventional Therapy (Placebo Comparator): Placebo was administered subcutaneously every 2 or 4 weeks over a period of 60 weeks to participants classified as having moderate to severe asthma. Doses (mg) and dosing frequency were determined by serum total IgE level (IU/mL) and body weight (kg). Also, participants continued with their conventional asthma therapy according to the National Asthma Education and Prevention Program (NAEPP-II, 2002) guidelines, under the management of an asthma specialist health care provider.
  Interventions: Biological: omalizumab placebo

INTERVENTIONS:
Biological: omalizumab — Subcutaneous injections of omalizumab will be administered every 2 or 4 weeks along with standard of care for asthma for 60 weeks, beginning with the Randomization Visit. Dosage is dependent on participant's individual characteristics.
  Other Names: Xolair®; Anti-IgE antibody,humanized monoclonal
  Arms: Omalizumab (Xolair) + Conventional Therapy
Biological: omalizumab placebo — Subcutaneous injections of placebo will be administered every 2 or 4 weeks along with standard of care for asthma for 60 weeks, beginning with the Randomization Visit. Dosage is dependent on participant's individual characteristics.
  Arms: Placebo + Conventional Therapy

SUMMARY:
The purpose of this study is to find out if adding omalizumab to standard asthma treatment results in a safer, more effective, and longer lasting asthma treatment strategy than standard treatment alone, in inner-city children with mild to severe asthma.

DETAILED DESCRIPTION:
This study is testing a medication called omalizumab for the treatment of asthma. Immunoglobulin E (IgE) is produced when one is exposed to allergens and it can cause inflammation in the lungs. Omalizumab can reduce inflammation and asthma attacks by blocking IgE. Unlike other medications for asthma, omalizumab is not an inhaler medication or pill. Instead, omalizumab is dissolved in a liquid and given by injection.

Studies indicate that people living in the inner-city areas are more likely to be exposed to indoor allergens that are difficult to avoid than people living in other areas. The purpose of this study is to find out if adding omalizumab to standard asthma treatment results in a safer, more effective, and longer lasting asthma treatment strategy than standard treatment alone.

This study will recruit inner-city children and adolescents with moderate to severe allergic asthma. This study will last about 1.5 to 2 years. Participants will be randomly assigned to receive either omalizumab or placebo injections once every 2 or 4 weeks. The injection schedule will be determined based on the participant's weight and total IgE. Both groups will receive standardized specialist care and basic asthma education including environmental control measures. Participants must have some form of health care insurance to cover the costs of asthma controller medications prescribed during the study.

Participants will complete a series of questionnaires about topics including perceived stress, home environment, physical activity, diet and nutrition, smoking habits, and quality of life. At study entry and monthly throughout the study, participants will complete questionnaires about their asthma symptoms and medical resource utilization. Some visits will include a physical examination, vital signs measurement, lung function tests, asthma medication evaluation, and an asthma action plan. Blood collection is required up to eight times during the study for safety labs.

ELIGIBILITY:
Inclusion Criteria:

* Both body weight and total serum IgE suitable for omalizumab dosing.
* Diagnosis of asthma made by a physician more than 1 year prior to study entry OR diagnosis of asthma made less than 1 year prior to study entry but have had asthma symptoms for longer than 1 year prior to study entry
* Are receiving long-term asthma control therapy OR have symptoms consistent with persistent asthma OR have evidence of uncontrolled disease
* Positive prick skin test to at least one perennial allergen (e.g., dust mite, cockroach, mold, cat, dog, rat, mouse)
* Live in a preselected zip code are
* Able to perform spirometry measurements
* Willing to sign informed consent or have parent or guardian willing to provide informed consent
* Previously had chicken pox or received varicella (chicken pox) vaccine
* Have some form of health care insurance that covers costs of medications

Exclusion Criteria:

If participant meets any of these criteria, they are not eligible at that time but may be reassessed:

* Systemic prednisone (or equivalent) during the 2 weeks prior to Visit 2
* Systemic prednisone (or equivalent) for more than 30 of the 60 days prior to study entry
* Pregnancy or breastfeeding
* Acute sinusitis or chest infection requiring antibiotics within 1 month of study screening
* Currently participating in another asthma-related clinical trial or have previously participated in an another asthma-related trial within 1 month of study entry
* Does not sleep at least 4 nights per week in one home
* Lives with a foster parent
* Does not have access to a phone
* Plans to move during the study
* Previously treated with anti-IgE therapy within 1 year of study entry
* Currently receiving or received hyposensitization therapy to any allergen in the year prior to study entry
* Previously received hyposensitization therapy to dust mite, Alternaria, or cockroach for more than 6 months in the 3 years prior to study entry

If participant meets any of these criteria, they are not eligible for the study and may not be reassessed:

* Significant medical illness. More information on this criterion can be found in the protocol.
* Certain medications within 4 weeks of study screening. More information on this criterion can be found in the protocol.
* Known hypersensitivity to any ingredients of omalizumab or related drugs
* Diagnosis of cancer, being investigated for possible cancer, or history of cancer
* Will not allow study physician to manage their asthma
* Does not primarily speak English (or Spanish at centers with Spanish-speaking staff)
* History of severe anaphylactoid or anaphylactic reaction(s)

Ages: 6 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 419 (Actual)
Dates: Start 2006-10; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William W. Busse, MD, Study Chair — University of Wisconsin, Madison; George T. O'Connor, MD, MS, Principal Investigator — Boston University; Jacqueline Pongracic, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago; Jamen Chmiel, MD, Principal Investigator — Rainbow Babies and Children's Hospital; Rebecca S. Gruchalla, MD, PhD, Principal Investigator — University of Texas Southwestern Medical Center; Andrew Liu, MD, Principal Investigator — National Jewish Health; Meyer Kattan, MD, CM, Principal Investigator — Columbia University; Wayne Morgan, MD, CM, Principal Investigator — University of Arizona Health Sciences Center; Stephen Teach, MD, MPH, Principal Investigator — Children's National Research Institute
Locations (8):
- United States (8):
  - University of Arizona Health Sciences Center, Tucson, Arizona
  - National Jewish Medical and Research Center, Denver, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Memorial Hospital, Chicago, Illinois
  - Boston University School of Medicine, Boston, Massachusetts
  - Columbia University Medical Center, New York, New York
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - University of Texas Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
Participant level data and additional relevant materials are available to the public in the Immunology Database and Analysis Portal (ImmPort). ImmPort is a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts.

REFERENCES:
- [Background] Ayres JG, Higgins B, Chilvers ER, Ayre G, Blogg M, Fox H. Efficacy and tolerability of anti-immunoglobulin E therapy with omalizumab in patients with poorly controlled (moderate-to-severe) allergic asthma. Allergy. 2004 Jul;59(7):701-8. doi: 10.1111/j.1398-9995.2004.00533.x. PMID 15180756
- [Background] Busse W, Corren J, Lanier BQ, McAlary M, Fowler-Taylor A, Cioppa GD, van As A, Gupta N. Omalizumab, anti-IgE recombinant humanized monoclonal antibody, for the treatment of severe allergic asthma. J Allergy Clin Immunol. 2001 Aug;108(2):184-90. doi: 10.1067/mai.2001.117880. PMID 11496232
- [Background] Mvula M, Larzelere M, Kraus M, Moisiewicz K, Morgan C, Pierce S, Post R, Nash T, Moore C. Prevalence of asthma and asthma-like symptoms in inner-city schoolchildren. J Asthma. 2005 Feb;42(1):9-16. doi: 10.1081/jas-200044746. PMID 15801322
- [Background] Szefler SJ, Apter A. Advances in pediatric and adult asthma. J Allergy Clin Immunol. 2005 Mar;115(3):470-7. doi: 10.1016/j.jaci.2004.12.1123. PMID 15753890
- [Result] Busse WW, Morgan WJ, Gergen PJ, Mitchell HE, Gern JE, Liu AH, Gruchalla RS, Kattan M, Teach SJ, Pongracic JA, Chmiel JF, Steinbach SF, Calatroni A, Togias A, Thompson KM, Szefler SJ, Sorkness CA. Randomized trial of omalizumab (anti-IgE) for asthma in inner-city children. N Engl J Med. 2011 Mar 17;364(11):1005-15. doi: 10.1056/NEJMoa1009705. PMID 21410369
- [Derived] Szefler SJ, Casale TB, Haselkorn T, Yoo B, Ortiz B, Kattan M, Busse WW. Treatment Benefit with Omalizumab in Children by Indicators of Asthma Severity. J Allergy Clin Immunol Pract. 2020 Sep;8(8):2673-2680.e3. doi: 10.1016/j.jaip.2020.03.033. Epub 2020 Apr 13. PMID 32298853
- See also: National Institute of Allergy and Infectious Diseases (NIAID) website — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) website — https://www.niaid.nih.gov/about/dait
- Available data/document: Individual Participant Data Set: SDY211 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY211 — ImmPort study identifier is SDY211.
- Available data/document: Study Protocol: SDY211 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY211 — ImmPort study identifier is SDY211.
- Available data/document: Study summary, -design, -adverse event(s), -interventions, -medications, -demographics, -study files.: SDY211 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY211 — ImmPort study identifier is SDY211.

RESULTS

PARTICIPANT FLOW:
Groups:
- Omalizumab (Xolair) + Conventional Therapy: Omalizumab was administered subcutaneously every 2 or 4 weeks over a period of 60 weeks to participants classified as having moderate to severe asthma. Doses (mg) and dosing frequency were determined by serum total immunoglobulin E (IgE) level (IU/mL) and body weight (kg). Also, participants continued with their conventional asthma therapy according to the National Asthma Education and Prevention Program (NAEPP-II, 2002) guidelines, under the management of an asthma specialist health care provider.
- Placebo + Conventional Therapy: Placebo was administered subcutaneously every 2 or 4 weeks over a period of 60 weeks to participants classified as having moderate to severe asthma. Doses (mg) and dosing frequency were determined by serum total immunoglobulin E (IgE) level (IU/mL) and body weight (kg). Also, participants continued with their conventional asthma therapy according to the National Asthma Education and Prevention Program (NAEPP-II, 2002) guidelines, under the management of an asthma specialist health care provider.
Period: Overall Study
Arm/Group | Omalizumab (Xolair) + Conventional Therapy | Placebo + Conventional Therapy
Started | 208 | 211
Completed | 155 | 157
Not Completed | 53 | 54

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Omalizumab (Xolair) + Conventional Therapy | Placebo + Conventional Therapy | Total
Number analyzed (Participants) | 208 | 211 | 419
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.9 (3.6) | 10.8 (3.4) | 10.8 (3.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 91 | 177
  Male | 122 | 120 | 242
Region of Enrollment [Number; unit: participants]
  United States | 208 | 211 | 419
Duration of Asthma at Baseline [Mean (Standard Deviation); unit: Years] — Asthma duration is the number of years since the participant was told by a physician that he/she has asthma, based upon the caretaker's response as reported at the baseline visit. This data was available for 332 of 419 (79%) study participants. Of the 332, 169 were from the Omalizumab (Xolair) + Conventional Therapy arm.
  Years | 7.5 (4.0) | 7.0 (3.8) | 7.3 (3.9)
Childhood Asthma Control Test (C-ACT) Score [Mean (Standard Deviation); unit: C-ACT score] — The Childhood Asthma Control Test (C-ACT) is a validated tool to assess overall asthma control (over the last 4 weeks) in patients ages 4 to 11 years. Scores can range from 0 to 27. A score of 19 or less is indicative of asthma that is not well controlled. The minimally important difference in C-ACT scores is not defined. C-ACT scores were available and relevant for 253 of 419 (60%) study participants. Of the 253, 123 were from the Omalizumab (Xolair) + Conventional Therapy arm.
  C-ACT score | 20.5 (3.8) | 20.7 (3.9) | 20.6 (3.8)
Asthma Control Test (ACT) Score [Mean (Standard Deviation); unit: ACT score] — The Asthma Control Test (ACT) is a validated tool to assess asthma control (over the last 4 weeks) in patients >= 12 yrs old. It is comprised of 5 questions assessing symptoms, use of rescue medications, and the impact of asthma on everyday functioning. All questions are scored on a 5-point Likert scale (higher score indicating better control). Total scores can range from 5-25. A score of <= 19 is indicative of not well-controlled asthma. The minimally important difference is 3 points. Scores were available for 166 of 419 participants (85 from the Omalizumab + Conventional Therapy arm).
  ACT score | 20.3 (3.8) | 20.3 (3.1) | 20.3 (3.5)
Maximum Number of Asthma Symptom Days (Previous 2 Weeks) [Mean (Standard Deviation); unit: Days] — Maximum symptom days was calculated as the largest of the following variables at the baseline visit: number of days with wheezing, chest tightness, or cough; number of nights of sleep disturbance; and number of days when activities were affected. This symptom scale ranges from 0 to 14 days per a 2-week look-back period. A higher score reflected a greater number of asthma symptoms.
  Days | 3.0 (3.5) | 3.1 (3.6) | 3.0 (3.5)
Missed Number of School Days (Previous 2 Weeks) [Mean (Standard Deviation); unit: Days] — The number of school days missed reported by the participant's caretaker was available for 339 of the 419 (81%) study participants. Of the 339, 164 were enrolled in the Omalizumab (Xolair) + Conventional Therapy arm.
  Days | 0.23 (0.76) | 0.25 (0.63) | 0.24 (0.70)
Forced Expiratory Volume in 1 Second (FEV1) % Predicted [Mean (Standard Deviation); unit: Percent] — FEV1 is air volume exhaled in 1 second during spirometry. For the trial, mild asthma is defined as pre-bronchodilator FEV1 ≥80% predicted, requiring no/low-moderate dose of inhaled glucocorticoids; moderate asthma and severe asthma, respectively, as pre-bronchodilator FEV1 <80% predicted requiring the same glucocorticoids as mild asthma and FEV1 <80% predicted requiring high-dose inhaled glucocorticoids (with/without continuous oral glucocorticoids) or uncontrolled despite treatment. FEV1 % of predicted is FEV1 converted to a percentage of normal, based on height, weight, and race.
  Percent | 93 (19) | 92 (18) | 93 (18)
FEV1/FVC Ratio [Mean (Standard Deviation); unit: ratio (x 100)] — The FEV1 (forced expiratory volume 1))/ FVC (forced vital capacity) ratio is used to evaluate airways obstructions since pure restrictive ventilatory defects cause an equal reduction in the FEV1 and the FVC. An FEV1/FVC ratio below 80% indicates airflow obstruction. Normal FEV1/FVC: 8 - 19 years of age=85%.
  Baseline FEV1/FVC ratio and FEV1 percent predicted data were available in 398 of the 419 participants. Of the 398, 204 were enrolled in the Omalizumab (Xolair) + Conventional Therapy arm.
  ratio (x 100) | 77.3 (10.0) | 77.6 (9.4) | 77.4 (9.7)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Number of Asthma Symptom Days
Description: Maximum symptom days was calculated as the largest of the following variables: number of days with wheezing, chest tightness, or cough; number of nights of sleep disturbance; and number of days when activities were affected. This symptom scale ranges from 0 to 14 days per a 2-week look-back period. A higher score reflected a greater number of asthma symptoms. Data represent an average of those collected in the time period (weeks 12-60), where at least one value was available in this assessment period and at baseline for a participant.
Time Frame: Weeks 12-60: 12 months of assessments starting 12 weeks after the initiation of study treatment.
Population: Intent-to-treat
Measure: Least Squares Mean (Standard Error); unit: Days
Arm/Group | Omalizumab (Xolair) + Conventional Therapy | Placebo + Conventional Therapy
Number analyzed (Participants) | 208 | 211
Days | 1.48 (0.10) | 1.96 (0.10)
Statistical Analysis 1: Comparison: Omalizumab (Xolair) + Conventional Therapy vs Placebo + Conventional Therapy; Maximum Symptom Day Comparison; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Linear mixed-effects models w/ random intercept and slope (to account for within-subject correlation over time) and visit and group as fixed effects

2. Secondary Outcome: Economic Outcome: Comparison of Number of Missed School Days Due to Asthma
Description: The number of school days missed was available for 307 of the 419 (73%) study participants, of which 152 were in the Omalizumab (Xolair) + Conventional Therapy arm. Source of data: caretaker/participant self-report. Data represent an average of those collected in the time period (weeks 12-60), where at least one value was available in this assessment period and at baseline for a participant.
Time Frame: Weeks 12-60: 12 months of assessments starting 12 weeks after the initiation of study treatment.
Population: Intent-to-treat
Measure: Least Squares Mean (Standard Error); unit: Days
Arm/Group | Omalizumab (Xolair) + Conventional Therapy | Placebo + Conventional Therapy
Number analyzed (Participants) | 152 | 155
Days | 0.16 (0.03) | 0.25 (0.03)
Statistical Analysis 1: Comparison: Omalizumab (Xolair) + Conventional Therapy vs Placebo + Conventional Therapy; Test type: Superiority or Other; p = 0.04, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: Economic Outcome: Number of Missed Work Days by Caretaker Due to Asthma
Description: The number of work days missed by the caretaker due to the study participant's asthma was available for 138 of 419 (33%) study participant caretakers. Source of data: caretaker self-report. Data represent an average of those collected in the time period (weeks 12-60).
Time Frame: Weeks 12-60: 12 months of assessments starting 12 weeks after the initiation of study treatment.
Population: Intent-to-treat
Measure: Least Squares Mean (Standard Error); unit: Days
Arm/Group | Omalizumab (Xolair) + Conventional Therapy | Placebo + Conventional Therapy
Number analyzed (Participants) | 69 | 69
Days | 0.13 (0.135) | 0.43 (0.121)
Statistical Analysis 1: Comparison: Omalizumab (Xolair) + Conventional Therapy vs Placebo + Conventional Therapy; Test type: Superiority or Other; p = 0.1111, Mixed Models Analysis; Linear mixed-effects models w/ random intercept (to account for within-subject correlation) and visit and group as fixed effects

4. Secondary Outcome: Child Asthma Control Test (C-ACT) Score
Description: The Childhood Asthma Control Test (C-ACT) is a validated tool to assess overall asthma control (over the last 4 weeks) in patients ages 4 to 11 years. Scores can range from 0 to 27. A score of 19 or less is indicative of asthma that is not well controlled. The minimally important difference in C-ACT scores is not defined. C-ACT scores were available as an outcome measure in 236 of the 419 participants, 118 of whom were in the Omalizumab (Xolair) + Conventional Therapy arm. Data represent an average of those collected in the time period (weeks 12-60), where at least one value was available in this assessment period and at baseline for a participant.
Time Frame: Weeks 12-60: 12 months of assessments starting 12 weeks after the initiation of treatment.
Population: Intent-to-treat
Measure: Least Squares Mean (Standard Error); unit: C-ACT score
Arm/Group | Omalizumab (Xolair) + Conventional Therapy | Placebo + Conventional Therapy
Number analyzed (Participants) | 118 | 118
C-ACT score | 23.0 (0.21) | 22.2 (0.21)
Statistical Analysis 1: Comparison: Omalizumab (Xolair) + Conventional Therapy vs Placebo + Conventional Therapy; Childhood Asthma Control Test comparison; Test type: Superiority or Other; p = 0.007, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]

5. Secondary Outcome: Asthma Control Test (ACT) Score
Description: The Asthma Control Test (ACT) is a validated tool to assess overall asthma control (over the last 4 weeks) in patients >= 12 years of age. It is a questionnaire comprised of 5 questions assessing: asthma symptoms, use of rescue medications, and the impact of asthma on everyday functioning. All questions are scored on a 5-point Likert scale, with a higher score indicating better control. All scores were added together to calculate a total score. Total scores can range from 5 to 25. A score of 19 or less is indicative of asthma that is not well controlled. The minimally important difference for ACT is 3 points. ACT scores as an outcome measure were available in 150 of the 419 participants, 77 of whom were in the Omalizumab (Xolair) + Conventional Therapy arm. Data represent an average of those collected in the time period (weeks 12-60), where at least one value was available in this assessment period and at baseline for a participant.
Time Frame: Weeks 12-60: 12 months of assessments starting 12 weeks after the initiation of study treatment.
Population: Intent-to-treat
Measure: Least Squares Mean (Standard Error); unit: ACT score
Arm/Group | Omalizumab (Xolair) + Conventional Therapy | Placebo + Conventional Therapy
Number analyzed (Participants) | 77 | 73
ACT score | 22.5 (0.22) | 22.3 (0.22)
Statistical Analysis 1: Comparison: Omalizumab (Xolair) + Conventional Therapy vs Placebo + Conventional Therapy; Asthma Control Test comparison; Test type: Superiority or Other; p = 0.54, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]

6. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) % Predicted
Description: FEV1 is air volume exhaled in 1 second during spirometry. For the trial, mild asthma is defined as pre-bronchodilator FEV1 ≥80% predicted, requiring no/low-moderate dose of inhaled glucocorticoids; moderate asthma and severe asthma, respectively, as pre-bronchodilator FEV1 <80% predicted requiring the same glucocorticoids as mild asthma and FEV1 <80% predicted requiring high-dose inhaled glucocorticoids (with/without continuous oral glucocorticoids) or uncontrolled despite treatment. FEV1 % of predicted is FEV1 converted to a percentage of normal, based on height, weight, and race. FEV1 percent predicted data as an outcome measure were available in 363 of the 419 participants, 190 of whom were in the Omalizumab (Xolair) + Conventional Therapy arm. Data represent an average of those collected in the time period (weeks 12-60), where at least one value was available in this assessment period and at baseline for a participant.
Time Frame: Weeks 12-60: 12 months of assessments starting 12 weeks after the initiation of study treatment.
Population: Intent-to-treat
Measure: Least Squares Mean (Standard Error); unit: Percent
Arm/Group | Omalizumab (Xolair) + Conventional Therapy | Placebo + Conventional Therapy
Number analyzed (Participants) | 190 | 173
Percent | 92.6 (0.60) | 91.7 (0.64)
Statistical Analysis 1: Comparison: Omalizumab (Xolair) + Conventional Therapy vs Placebo + Conventional Therapy; FEV1 % of predicted value comparison; Test type: Superiority or Other; p = 0.30, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]

7. Secondary Outcome: FEV1/FVC Ratio
Description: The FEV1 (forced expiratory volume 1))/ FVC (forced vital capacity) ratio is used to evaluate airways obstructions since pure restrictive ventilatory defects cause an equal reduction in the FEV1 and the FVC. An FEV1/FVC ratio below 80% indicates airflow obstruction. Normal FEV1/FVC: 8 - 19 years of age=85%.
  FEV1/FVC ratio data as an outcome measure were available in 363 of the 419 participants, 190 of whom were in the Omalizumab (Xolair) + Conventional Therapy arm. Data represent an average of those collected in the time period (weeks 12-60), where at least one value was available in this assessment period and at baseline for a participant.
Time Frame: Weeks 12-60: 12 months of assessments starting 12 weeks after the initiation of study treatment.
Population: Intent-to-treat
Measure: Least Squares Mean (Standard Error); unit: Ratio (x100)
Arm/Group | Omalizumab (Xolair) + Conventional Therapy | Placebo + Conventional Therapy
Number analyzed (Participants) | 190 | 173
Ratio (x100) | 77.3 (0.36) | 77.5 (0.38)
Statistical Analysis 1: Comparison: Omalizumab (Xolair) + Conventional Therapy vs Placebo + Conventional Therapy; FEV1:FVC ×100 comparison; Test type: Superiority or Other; p = 0.81, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]

8. Secondary Outcome: Exhaled Nitric Oxide
Description: Exhaled nitric oxide is a biomarker of airway inflammation. Measurement (in parts per billion,ppb) of exhaled nitric oxide (eNO) prior to spirometry, employing a technique modified after Silkoff et al (1997) and following American Thoracic Society guidelines for eNO assessment (American Thoracic Society, 1999). Nitric oxide concentrations were measured using a rapid-response chemiluminescent analyzer (NIOX™ System, Aerocrine, Sweden) which has a response time of < 700 ms for 10-90% full scale. The Food and Drug Administration has approved this device for clinical application in asthma management. Data represent an average of those collected in the time period (weeks 12-60), where at least one value was available in this assessment period and at baseline for a participant.
Time Frame: Weeks 12-60: 12 months of assessments starting 12 weeks after the initiation of study treatment.
Population: Intent-to-treat
Measure: Least Squares Mean (Standard Error); unit: ppb
Arm/Group | Omalizumab (Xolair) + Conventional Therapy | Placebo + Conventional Therapy
Number analyzed (Participants) | 152 | 145
ppb | 22.6 (1.46) | 33.0 (1.50)
Statistical Analysis 1: Comparison: Omalizumab (Xolair) + Conventional Therapy vs Placebo + Conventional Therapy; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]

9. Secondary Outcome: Percent Adherence to Asthma Medication
Description: Adherence to the study regimen and other asthma treatments, assessed as percent of expected dose taken, by means of study interviews and study physician corroboration every 3 months. Adherence data as an outcome were available in 384 of the 419 participants, 193 of whom were in the Omalizumab (Xolair) + Conventional Therapy arm. Data represent an average of those collected in the time period (weeks 12-60), where at least one value was available in this assessment period and at baseline for a participant.
Time Frame: Weeks 12-60: 12 months of assessments starting 12 weeks after the initiation of study treatment
Population: Intent-to-treat
Measure: Least Squares Mean (Standard Error); unit: percentage of expected dose taken
Arm/Group | Omalizumab (Xolair) + Conventional Therapy | Placebo + Conventional Therapy
Number analyzed (Participants) | 193 | 191
percentage of expected dose taken | 84.6 (1.78) | 88.6 (1.80)
Statistical Analysis 1: Comparison: Omalizumab (Xolair) + Conventional Therapy vs Placebo + Conventional Therapy; Percent Adherence Comparison; Test type: Superiority or Other; p = 0.12, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]

10. Secondary Outcome: Percent Prevalence: Treatment Step Level 1 or 2 (Mild Asthma)
Description: Treatment steps were established, per the National Asthma Education and Prevention Program Expert Panel Report 3 guidelines. Steps 1-2 apply to mild asthma, 3 to moderate asthma, and 4-6 to severe asthma. At Step 0, the recommendation is for no asthma-control medication or albuterol as needed; at 1, budesonide 180 mcg once a day; at 2, budesonide 180 mcg twice a day; at 3, budesonide 360 mcg twice a day; at 4, fluticasone-salmeterol (Advair, GlaxoSmithKline) 250 mcg fluticasone and 50 mcg salmeterol twice a day; at 5, Advair 250 mcg and 50 mcg twice a day plus montelukast once a day; and at 6, Advair 500 mcg and 50 mcg twice a day plus montelukast once a day. (The doses for montelukast are 5 mg per day for those <=14 years old and 10 mg per day for those >=15 years.) Data represent an average of those in the time period, where at >/= 1 value was available in this period and at baseline for a participant; results are model predicted numbers (e.g.,odds ratios converted to percentages).
Time Frame: Weeks 12-60: 12 months of assessments starting 12 weeks after the initiation of study treatment
Population: Intent-to-treat
Measure: Number; unit: percent prevalence
Arm/Group | Omalizumab (Xolair) + Conventional Therapy | Placebo + Conventional Therapy
Number analyzed (Participants) | 208 | 211
percent prevalence | 43.6 (4.0) | 26.7 (3.3)
Statistical Analysis 1: Comparison: Omalizumab (Xolair) + Conventional Therapy vs Placebo + Conventional Therapy; Step level 1- 2 (mild asthma) Percent Comparison; Test type: Superiority or Other; p = 0.001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]

11. Secondary Outcome: Percent Prevalence: Treatment Step Level 4 Through 6 (Severe Asthma)
Description: Steps were established, per the National Asthma Education and Prevention Program Expert Panel Report 3 guidelines. Steps 1-2 apply to mild asthma, 3 to moderate asthma, and 4-6 to severe asthma. At Step 0, the recommendation is for no asthma-control medication or albuterol as needed; at 1, budesonide 180 mcg once a day; at 2, budesonide 180 mcg twice a day; at 3, budesonide 360 mcg twice a day; at 4, fluticasone-salmeterol (Advair, GlaxoSmithKline) 250 mcg fluticasone and 50 mcg salmeterol twice a day; at 5, Advair 250 mcg and 50 mcg twice a day plus montelukast once a day; and at 6, Advair 500 mcg and 50 mcg twice a day plus montelukast once a day. (The doses for montelukast are 5 mg per day for those <=14 years old and 10 mg per day for those >=15 years.) Data represent an average of those in the time period, where at least one value was available in this period and at baseline for a participant. Results values are model predicted numbers,(e.g, odds ratios converted to percentages).
Time Frame: Weeks 12-60: 12 months of assessments starting 12 weeks after the initiation of study treatment
Population: Intent-to-treat
Measure: Number; unit: percent prevalence
Arm/Group | Omalizumab (Xolair) + Conventional Therapy | Placebo + Conventional Therapy
Number analyzed (Participants) | 208 | 211
percent prevalence | 31.2 (3.5) | 50.8 (4.0)
Statistical Analysis 1: Comparison: Omalizumab (Xolair) + Conventional Therapy vs Placebo + Conventional Therapy; Step level 4 - 6 (severe asthma)percent comparison; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]

12. Secondary Outcome: Dose Inhaled Corticosteroids (Glucocorticoids)
Description: Prescribed dose (mcg/day) of inhaled glucocorticoids to maintain asthma control. The dose of inhaled glucocorticoids was converted to the budesonide-equivalent dose. Data represent an average of those collected in the time period (weeks 12-60), where at least one value was available in this assessment period and at baseline for a participant.
Time Frame: Weeks 12-60: 12 months of assessments starting 12 weeks after the initiation of study treatment.
Population: Intent-to-treat
Measure: Least Squares Mean (Standard Error); unit: mcg/day
Arm/Group | Omalizumab (Xolair) + Conventional Therapy | Placebo + Conventional Therapy
Number analyzed (Participants) | 208 | 211
mcg/day | 663 (23.3) | 771 (23.5)
Statistical Analysis 1: Comparison: Omalizumab (Xolair) + Conventional Therapy vs Placebo + Conventional Therapy; Inhaled glucocorticoids prescribed - mcg per day comparison; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]

13. Secondary Outcome: Percent Prevalence: Prescribed Rescue Beta 2 Agonists
Description: Percent of participants prescribed long-acting beta 2 agonists to maintain asthma control. Data represent an average of those collected in the time period (weeks 12-60), where at least one value was available in this assessment period and at baseline for a participant. Results values are model predicted numbers, (e.g.,odds ratios converted to percentages).
Time Frame: Weeks 12-60: 12 months of assessments starting 12 weeks after the initiation of study treatment.
Population: Intent-to-treat
Measure: Number; unit: percent prevalence
Arm/Group | Omalizumab (Xolair) + Conventional Therapy | Placebo + Conventional Therapy
Number analyzed (Participants) | 208 | 211
percent prevalence | 55.4 (2.4) | 65.5 (2.5)
Statistical Analysis 1: Comparison: Omalizumab (Xolair) + Conventional Therapy vs Placebo + Conventional Therapy; Comparison percent prescribed long-acting beta 2 agonists; Test type: Superiority or Other; p = 0.003, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]

14. Secondary Outcome: Percent Prevalence: Asthma-Related Medical Care Resource Utilization - Hospitalizations
Description: Percent participants with >=1 hospitalizations. A hospitalization is defined as an asthma-related, overnight hospitalization. . Results values are model predicted numbers,(e.g., odds ratios converted to percentages).
Time Frame: Weeks 12-60: 12 months of assessments starting 12 weeks after the initiation of study treatment.
Population: Intent-to-treat
Measure: Number; unit: percent prevalence
Arm/Group | Omalizumab (Xolair) + Conventional Therapy | Placebo + Conventional Therapy
Number analyzed (Participants) | 208 | 211
percent prevalence | 1.5 (0.9) | 6.3 (1.8)
Statistical Analysis 1: Comparison: Omalizumab (Xolair) + Conventional Therapy vs Placebo + Conventional Therapy; Test type: Superiority or Other; p = 0.02, Regression, Logistic; Hospitalizations were summed over the course of the double-blind & analyzed with logistic regression (LR) of 'any' vs. 'none'. The LR was unadjusted

15. Secondary Outcome: Percent Prevalence: Asthma Exacerbations
Description: Percent participants with >=1 exacerbations. An exacerbation was defined as a prednisone burst (a minimum of 20 mg per day of prednisone, or the equivalent, taken for any 3 of 5 consecutive days) or hospitalization. Results values are model predicted numbers, (e.g.,odds ratios converted to percentages).
Time Frame: Weeks 12-60: 12 months of assessments starting 12 weeks after the initiation of study treatment.
Population: Intent-to-treat
Measure: Number; unit: percent prevalence
Arm/Group | Omalizumab (Xolair) + Conventional Therapy | Placebo + Conventional Therapy
Number analyzed (Participants) | 208 | 211
percent prevalence | 30.3 (3.3) | 48.8 (3.7)
Statistical Analysis 1: Comparison: Omalizumab (Xolair) + Conventional Therapy vs Placebo + Conventional Therapy; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Exacerbations were summed over the course of the double-blind and analyzed with an LR of 'any' versus 'none'. LR adjusted for study site and dosing

16. Secondary Outcome: Asthma Caregiver's Quality of Life Questionnaire (PACQLQ) Overall Score
Description: Asthma-Specific Quality of Life (QOL) Measure . The PACQLQ is a validated tool that measures limitations and anxieties faced by primary caregivers of children with asthma. Scores are calculated as the mean score within two domains of questions (re: activity limitation and emotional function) and overall scores represent the mean across all questions. The use of the PACQLQ is valid for use in the caretakers of children ages 7 to 17 years of age. Higher scores indicate better quality of life. Minimum possible score is 1 (maximum impairment); maximum possible score is 7 (no impairment). The range of actual scores were a minimum of 2.4 and a maximum of 7.
  Method: Caretaker self-report. PACQLQ scores were available for 320 of 419 (76%) of study participant caretakers (159 in the Omalizumab (Xolair) + Conventional Therapy arm).
Time Frame: Week 60
Population: Intent-to-treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Omalizumab (Xolair) + Conventional Therapy | Placebo + Conventional Therapy
Number analyzed (Participants) | 159 | 161
units on a scale | 5.7 (1.2) | 5.8 (1.1)
Statistical Analysis 1: Comparison: Omalizumab (Xolair) + Conventional Therapy vs Placebo + Conventional Therapy; Test type: Superiority or Other; p = 0.84, Wilcoxon (Mann-Whitney)

17. Secondary Outcome: Paediatric Asthma Quality of Life Questionnaire (PAQLQ) Overall Score
Description: Asthma-specific quality of life (QOL) validated tool designed for children 7 to 17 years of age. PAQLQ measures functional problems that are most troublesome to children with asthma. PAQLQ has 23 questions in 3 domains (activity limitation=5, emotional function=8, symptoms=10). Patients responded to each question on a 7-point Likert scale. Overall PAQLQ score is mean of 23 questions; each domain score is mean of questions in that domain. Minimum possible score is 1 (maximum impairment); maximum possible score is 7 (no impairment). Actual scores ranged from 2.1 to 7.
  PAQLQ scores were available for 338 of 419 (81%) of study participants, 170 of whom were in the Omalizumab (Xolair) + Conventional Therapy arm.
Time Frame: Week 60
Population: Intent-to-treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Omalizumab (Xolair) + Conventional Therapy | Placebo + Conventional Therapy
Number analyzed (Participants) | 170 | 168
units on a scale | 6.1 (1.0) | 6.2 (0.9)
Statistical Analysis 1: Comparison: Omalizumab (Xolair) + Conventional Therapy vs Placebo + Conventional Therapy; Test type: Superiority or Other; p = 0.58, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Omalizumab (Xolair) + Conventional Therapy | Placebo + Conventional Therapy
Serious Adverse Events (participants affected / at risk) | 24/208 | 34/211
Other Adverse Events (participants affected / at risk) | 32/208 | 32/211
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omalizumab (Xolair) + Conventional Therapy (N=208) | Placebo + Conventional Therapy (N=211)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 4 (4)
Food allergy (Immune system disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Burns second degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Diabetes mellitus insulin-dependent (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Intra-uterine death (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Affective disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Aggression (Psychiatric disorders) | 1 (1) | 1 (1)
Anger (Psychiatric disorders) | 0 (0) | 1 (1)
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Genital disorder female (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 13 (17) | 20 (24)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Tonsillar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omalizumab (Xolair) + Conventional Therapy (N=208) | Placebo + Conventional Therapy (N=211)
Respiratory tract infection (Infections and infestations) | 14 (27) | 18 (34)
Upper respiratory tract infection (Infections and infestations) | 19 (25) | 20 (34)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No